CLINICAL TRIAL: NCT00005675
Title: Multicenter Phase II Trial of Oral Type I Bovine Collagen in Scleroderma
Brief Title: Oral Type I Collagen for Relieving Scleroderma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Collaborators: Wayne State University (Other); University of California, Los Angeles (Other); UTHSC (Unknown); Medical University of South Carolina (Other); Beth Israel Medical Center (Other); University of Alabama at Birmingham (Other); Johns Hopkins University (Other); Georgetown University (Other); Baltimore VA Medical Center (U.S. Federal Agency); Northwestern University (Other)
Responsible Party: Arnold E. Postlethwaite, MD, UTHSC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01 AR92242; NIAMS-048
Expanded Access: Available
Record Dates: First submitted 2000-05-26; First posted 2000-05-29 (Estimated); Last update posted 2010-05-25 (Estimated); Status verified 2008-03

CONDITIONS: Scleroderma; Connective Tissue Diseases
Keywords: Systemic Scleroderma (SSc); Bovine Type I Collagen (CI); Multicenter
MeSH Terms: conditions — Scleroderma, Diffuse; Connective Tissue Diseases; Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive oral bovine type I collagen (CI) daily for 15 months
  Interventions: Drug: Oral bovine type I collagen
- 2 (Placebo Comparator): Participants will receive placebo daily for 15 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral bovine type I collagen — 500 mcg of CI daily for 15 months
  Other Names: CI
  Arms: 1
Drug: Placebo — CI placebo daily for 15 months
  Arms: 2

SUMMARY:
Diffuse systemic sclerosis (SSc), or scleroderma, is a connective tissue disease causing damage to skin and other organs. The purpose of this study is to determine if taking oral bovine type I collagen (CI) will improve the condition of SSc patients.

DETAILED DESCRIPTION:
SSc is a chronic connective tissue disease that is caused by excess collagen deposits that damage the skin and other organs. This study will determine if a daily oral dose of bovine CI will improve the condition of patients with SSc.

Patients will be randomly assigned to one of two groups. The first group will receive 500 mcg bovine CI daily for 15 months; the second group will receive placebo. Study visits will be conducted at Months 4, 8, 12, and 15. Patients will undergo physical examination and blood tests at each visit. Patients will also be evaluated for modified Rodnan skin score (MRSS) and will be given health assessment questionnaires. A chest x-ray will be conducted at study entry and pulmonary function tests will be conducted at study entry and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diffuse systemic scleroderma (by American College of Rheumatology criteria 1980) of 10 years or less
* Stable skin involvement by history or physical examination 6 months prior to study entry
* Stable modified Rodnan skin score (MRSS) for 1 month prior to study entry
* Stable MRSS of 16 or more at screening and stable MRSS between screening and baseline visit
* Agree to use acceptable forms of contraception

Exclusion Criteria:

* Participation in another clinical research study involving evaluation of another investigational drug within 90 days prior to study entry
* Concurrent serious medical condition which, in the opinion of the investigator, makes the patient inappropriate for the study
* Systemic sclerosis-like illnesses associated with environmental, ingested, or injected agents, such as L-tryptophan, tainted rapeseed oil, vinyl chloride, or bleomycin
* Limited and localized (morphea) or linear SSc
* Tenderness or swelling of the extremities (eosinophilic fasciitis)
* Pregnancy
* Use of certain medications
* Allergy to beef or dairy products
* Nonsteroidal anti-inflammatory drugs (NSAIDs) within 1 week before baseline visit. Aspirin at 325 mg or less daily for stroke or heart attack prevention is allowed.
* Use of herbal and some alternative therapies
* Any organ transplant or stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2000-04; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Disease condition, as measured by physical exam, modified Rodnan skin score (MRSS), health assessment questionnaires, chest x-ray, and pulmonary function tests | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Arnold E. Postlethwaite, MD, Principal Investigator — University of Tennessee at Memphis
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University School Of Medicine, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Beth Israel Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Virginia Mason Research Center, Seattle, Washington

REFERENCES:
- [Background] Postlethwaite AE. Can we induce tolerance in rheumatoid arthritis? Curr Rheumatol Rep. 2001 Feb;3(1):64-9. doi: 10.1007/s11926-001-0052-z. PMID 11177772
- [Background] Carbone LD, McKown K, Pugazhenthi M, Barrow KD, Warrington K, Somes G, Postlethwaite AE. Dosage effects of orally administered bovine type I collagen on immune function in patients with systemic sclerosis. Arthritis Rheum. 2004 Aug;50(8):2713-5. doi: 10.1002/art.20361. No abstract available. PMID 15334493
- [Derived] Postlethwaite AE, Wong WK, Clements P, Chatterjee S, Fessler BJ, Kang AH, Korn J, Mayes M, Merkel PA, Molitor JA, Moreland L, Rothfield N, Simms RW, Smith EA, Spiera R, Steen V, Warrington K, White B, Wigley F, Furst DE. A multicenter, randomized, double-blind, placebo-controlled trial of oral type I collagen treatment in patients with diffuse cutaneous systemic sclerosis: I. oral type I collagen does not improve skin in all patients, but may improve skin in late-phase disease. Arthritis Rheum. 2008 Jun;58(6):1810-22. doi: 10.1002/art.23501. PMID 18512816